CLINICAL TRIAL: NCT05498116
Title: Effect of Montelukast on Kidney and Vascular Function in Type 1 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-1027
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Albuminuria
MeSH Terms: conditions — Albuminuria | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): One capsule daily
  Interventions: Other: Placebo
- Montelukast (Experimental): One 10mg capsule daily
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — 10mg daily
  Arms: Montelukast
Other: Placebo — 1 capsule daily
  Arms: Placebo

SUMMARY:
Kidney disease is a common problem among people with type 1 diabetes and can lead to disability, dialysis, and early death. Inflammation plays a key role in the development of kidney disease in type 1 diabetes and targeting leukotrienes, inflammatory chemicals the body releases in response to allergic reactions, may represent a promising therapy to slow the progression of diabetic kidney disease. The current proposal will investigate whether montelukast, a leukotriene blocker, lowers increased levels of protein in the urine (an early marker of diabetic kidney disease), and improves kidney and cardiovascular function in people with type 1 diabetes and kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Type 1 diabetes for at least 5 years
* Urine albumin to creatinine ratio 30-5000 mg/g on first morning void
* eGFR 30-89 ml/min/1.73m2 at time of screening
* Blood pressure <140/90 mm Hg prior to randomization
* Use of angiotensin converting enzyme inhibitor or angiotensin receptor blocker with stable dose for 4 weeks
* BMI < 40 kg/m2 (FMDBA measurements can be inaccurate in severely obese patients).
* Stable anti-hypertensive regimen for at least one month prior to randomization
* Stable regimen of insulin delivery, i.e. automated insulin delivery (AID) system or multiple daily injections) 4 weeks prior to randomization
* Sedentary or recreationally active (≤2 days of vigorous aerobic exercise as vigorous exercise may affect vascular function measurements)
* Able to provide consent

Exclusion Criteria:

* Significant comorbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Uncontrolled hypertension
* Factors judged to limit adherence to interventions
* Anticipated initiation of dialysis or kidney transplantation within 6 months
* Current participation in another research study
* Pregnancy or planning to become pregnant or currently breastfeeding
* Allergy to aspirin
* Severe hepatic impairment (Child-Pugh Class C)
* History of major psychiatric disorder
* Use of inhaled or systemic corticosteroids or long-acting beta agonists (higher risk of neuropsychiatric reaction)
* Penicillin allergy
* Iodine allergy
* Shellfish allergy
* Current use of phenobarbital, rifampin or carbamazepine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Albuminuria | Baseline, 6 months
  Change in albuminuria from baseline to 6 months

SECONDARY OUTCOMES:
Change in Brachial artery flow mediated dilation (FMD) | Baseline, 6 months
  Change in FMD from baseline to 6 months
Change in Large Elastic Artery Stiffness | Baseline, 6 months
  Change in aortic pulse wave velocity from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No